CLINICAL TRIAL: NCT03263065
Title: A Pilot Participant-blind Study of the Effect of Bran, Psyllium and Nopal on Intestinal Water Content Using Magnetic Resonance Imaging
Brief Title: A Study of the Effect of Bran, Psyllium and Nopal on Intestinal Water Content Using Magnetic Resonance Imaging
Acronym: NOPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NOPAL
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-05

CONDITIONS: Constipation; Diet Modification
Keywords: Nopal; Bran; Psyllium
MeSH Terms: conditions — Constipation | interventions — Psyllium

STUDY DESIGN:
Intervention Model Description: This will be a three-period, three-treatment crossover trial with blinding of data analysis
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nopal added to test meal (Experimental): test meal including nopal powder
  Interventions: Dietary Supplement: Nopal
- Psyllium added to test meal (Experimental): test meal including psyllium powder
  Interventions: Dietary Supplement: Psyllium
- Bran added to test meal (Experimental): test meal including bran powder
  Interventions: Dietary Supplement: Bran

INTERVENTIONS:
Dietary Supplement: Bran — 220g rice pudding meal with raspberry jam with added bran flakes
  Arms: Bran added to test meal
Dietary Supplement: Nopal — 220g rice pudding meal with raspberry jam with added nopal flakes
  Arms: Nopal added to test meal
Dietary Supplement: Psyllium — 220g rice pudding meal with raspberry jam with added psyllium flakes
  Arms: Psyllium added to test meal

SUMMARY:
This study will compare 3 food products (bran, psyllium and nopal) on intestinal water content measured via MRI.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The role of dietary fibre in human health is a topic of both debate and research. Interpreting evidence is complicated by changes in the definition of fibre. In the UK the Scientific Advisory Committee for Nutrition has recently proposed a definition of "all carbohydrates that are neither digested nor absorbed in the small intestine and have a degree of polymerisation of three or more monomeric units, plus lignin". They have also called for further research into the physiological effects of fibre of the gastrointestinal (GI) tract.

The Nottingham GI MRI group has been at the forefront of elucidating the effects of poorly digested carbohydrates on gastrointestinal physiology. The investigators have published techniques to measure free water in the small bowel and assessment of the physical form of chyme in the colon using MR relaxometry. This includes the demonstration that fructose ingestion on its own leads to increased free water in the small bowel compared to co-ingestion with glucose.

Bran is often confused with dietary fibre. Although it contains fibre, the term actually refers to the outer husk of seeds and grains. It has been shown to accelerate oro-caecal transit (OCT) with scintigraphy. Bran can also be shown to increase small bowel water content, possibly by mechanical stimulation, one of the most powerful stimuli for small intestinal secretion, which may be a mechanism to prevent blockage. In the past bran's high fibre content led to the hypothesis that its effect derived from holding water in the lumen but a comparison study of 17 different fibres found an inverse relationship between their water-holding properties and effect on faecal weight, with bran holding the least water but inducing the largest weight changes. Rather, weight change appeared to relate to the amount of undigested fibre present in the faeces and the associated changes in bacterial numbers, which account for most of dry stool weight.

In contrast, psyllium husk contains a fibre that binds water effectively. On this basis it has been used as a laxative for thousands of years. In fact, there is little evidence that psyllium accelerates whole gut transit time as might be expected of a laxative. Work within the investigating group has shown that psyllium increases water in both the small bowel and the faeces, leading to softer, looser stool.

Nopal is a Mexican dietary product derived from cactus. It contains a different mix of fibre, 2/3rds of which is insoluble like bran fibre and 1/3rd soluble like psyllium. It is the subject of several health claims. The investigating group has recently been awarded a grant by the Newton Fund, through the Medical Research council, to study its effects on gut function. The aim of the Newton Fund is to stimulate collaborative research with middle-income countries such as Mexico. Part of the project plan is to invite a Mexican radiologist, Dr Alfonso Gil-Valadez, to Nottingham to learn about the MRI techniques used by our group.

TRIAL OBJECTIVES AND PURPOSE

Purpose

The purpose of the study is to gather pilot data on the effect of Nopal on intestinal water content, in comparison to bran and psyllium.

Objective

The primary objective is to gather pilot data on the change from baseline in small bowel water content in healthy volunteers after a meal containing nopal, in comparison to meals containing psyllium or bran.

Secondary Objectives

Secondary objectives will be to gather pilot data on the effects of the fibre-containing meals on the physical form of colonic chyme, colonic volume and breath markers of fermentation.

Hypotheses

The test meals will lead to differences in post-prandial water in the small bowel.

The test meals will lead to differences in the post-prandial volume and physical composition of chyme in the colon.

The test meals will not lead to change in breath markers of fermentation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Able to give informed consent

Exclusion Criteria:

* Pregnancy declared by candidate
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function
* A positive diagnosis of irritable bowel syndrome based on the Rome IV criteria questionnaire
* Reported history of previous resection of the oesophagus, stomach or intestine (excluding appendix)
* Intestinal stoma
* Any medical condition making participation potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner, known allergy to one of the food products
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Will not agree to dietary restrictions required in 24 hours before each MRI study day
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM
* Participation in any medical trials for the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in T1 relaxation time (ms) of the chyme in the ascending colon | baseline, immediately post ingestion, 1, 2, 3 and 4 hours post ingestion
  measured by MRI

SECONDARY OUTCOMES:
Change from the baseline in small bowel water content (mL) | baseline, immediately post ingestion, 1, 2, 3 and 4 hours post ingestion
  measured by MRI
Change from the baseline in colonic volume in mL | baseline, immediately post ingestion, 1, 2, 3 and 4 hours post ingestion
  measured by MRI
Change from the baseline of breath hydrogen and methane (ppm) | baseline, immediately post ingestion, 1, 2, 3 and 4 hours post ingestion
  measured using GastroCHeck

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, PhD, Study Chair — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunn D, Murthy R, Major G, Wilkinson-Smith V, Hoad C, Marciani L, Remes-Troche J, Gill S, Rossi M, Harris H, Ahn-Jarvis J, Warren F, Whelan K, Spiller R. Contrasting effects of viscous and particulate fibers on colonic fermentation in vitro and in vivo, and their impact on intestinal water studied by MRI in a randomized trial. Am J Clin Nutr. 2020 Sep 1;112(3):595-602. doi: 10.1093/ajcn/nqaa173. PMID 32619212